CLINICAL TRIAL: NCT05535192
Title: TeleHealth Resistance Exercise Intervention to Preserve Dose Intensity and Vitality in Elder Breast Cancer Patients (THRIVE-65)
Brief Title: TeleHealth Resistance Exercise Intervention to Preserve Dose Intensity and Vitality in Elder Breast Cancer Patients
Acronym: THRIVE-65
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Case Western Reserve University (Other); University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jennifer A. Ligibel, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-250; 1U01CA271277-01 (NIH)
Record Dates: First submitted 2022-08-29; First posted 2022-09-10 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer; Stage III Breast Cancer; Breast Cancer Female; Stage I Breast Cancer; Stage II Breast Cancer
Keywords: Breast Cancer; Stage III Breast Cancer; Stage II Breast Cancer; Stage I Breast Cancer; Exercise Intervention; Nutrition Intervention; Supportive Care
MeSH Terms: conditions — Breast Neoplasms | interventions — Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HEALTH EDUCATION AND SUPPORT CONTROL GROUP (Active Comparator): The research study procedures include screening for eligibility and a baseline visit to collect measurements and questionnaires. After the baseline appointment, participants randomized into the Heath Education Support Program will receive a tablet from the study that is pre-loaded with material to help support them during chemotherapy. The tablet materials will include supportive care and resources that focus on movement (light stretching and gentle yoga), soothing music, meditation/mindfulness, and recipes/cooking demos. Participants in this arm will be asked to fill out questionnaires at the start of each chemotherapy cycle to indicate any side effects from chemotherapy and the amount of time they spend engaging with the tablet. At the end of participants' chemotherapy, they will be asked to complete end-of-study measures.
  Interventions: Behavioral: Health Education Support Program
- THRIVE: EXERCISE INTERVENTION WITH PROTEIN INTAKE SUPPORT (Experimental): The research study procedures include screening for eligibility and a baseline visit to collect measurements and questionnaires. After the baseline appointment, participants randomized into the THRIVE Exercise and Diet Intervention will work with a coach to gradually build exercise and stay active during chemotherapy treatment. Participants will work with an exercise coach to reach the muscle strengthening and aerobic exercise goals of the study. Participants will also consult with a dietician to ensure adequate protein intake during the study. Participants in this arm will be asked to fill out questionnaires at the start of each chemotherapy cycle to indicate any side effects from chemotherapy. At the end of participants' chemotherapy, they will be asked to complete end-of-study measures.
  Interventions: Behavioral: THRIVE

INTERVENTIONS:
Behavioral: THRIVE — The THRIVE Intervention will involve:
  1) one in-person exercise sessions, followed by twice-weekly, home-based exercise sessions, supervised remotely through telehealth, and 2) a remotely delivered dietary assessment and recommendations to support protein intake throughout the study
  Arms: THRIVE: EXERCISE INTERVENTION WITH PROTEIN INTAKE SUPPORT
Behavioral: Health Education Support Program — Participants will receive a tablet with information and resources regarding mediation, stretching and gentle movement, relaxation and creative arts during chemotherapy
  Arms: HEALTH EDUCATION AND SUPPORT CONTROL GROUP

SUMMARY:
This research is being done to assess whether an exercise intervention with protein intake support vs a health education and support program will make it easier for women age 65 or older who are receiving chemotherapy for breast cancer to receive all of their planned chemotherapy according to schedule and at the planned dose.

DETAILED DESCRIPTION:
The research study procedures include screening for eligibility. After participants are determined to be eligible and have signed consent, they will participate in a baseline visit to collect measurements (e.g., weight/height/waist measurements) and questionnaires, a memory test, functional movement and strength testing, and a physical activity assessment. After baseline measures are collected, participants will be randomized to either the THRIVE Exercise and Diet Intervention or the Heath Education and Support Program during chemotherapy. There is a follow up visit up to 4 weeks after the completion of chemotherapy to repeat measurements and questionnaires.

The duration of the study will be 10-26 weeks, depending on the type of chemotherapy participants are receiving.

The THRIVE Intervention will involve:

* Exercise: Participants in the THRIVE Intervention arm work with an exercise coach to participate in both muscle strengthening exercises and aerobic exercises. There is one in-person exercise session at the beginning of the study. The remainder of the exercise sessions are done twice weekly via telehealth throughout chemotherapy treatment.
* Protein intake support: Participants in the THRIVE Intervention will meet with a dietitian to make sure they are eating enough protein throughout their chemotherapy treatments. Participants will be asked to keep a daily protein checklist and share this with the exercise coach each week.

The Health Education Support Program will involve:

- Health education tablet: Participants in the Health Education Support program will receive a tablet with information regarding mediation, stretching and gentle movement, relaxation and creative arts throughout chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Women age >=65
* Diagnosed with stage I-III invasive breast cancer
* BMI between 18-50 kg/m2
* Scheduled to begin at least 10 weeks of neoadjuvant or adjuvant cytotoxic chemotherapy for curative intent
* If enrolled in clinical chemotherapy drug trial, considered eligible if regimen includes an anthracycline or a taxane, unless the trial alters the chemotherapy agents/doses according to patient response (e.g.; I-SPY trials)
* Self-reported ability to walk for 6 minutes and/or 2 blocks (with or without assistive device)
* Ability to provide written informed consent.
* Ability to understand, speak, and read English. This is because many of the study instruments used are not readily available in multiple languages. Additionally, site-based study staff, such as exercise physiologists, are not bilingual and not all sites have access to interpreters.

Exclusion Criteria:

* Following a therapeutic diet for co-morbid disease where the THRIVE-65 diet would be contraindicated as assessed by the RD
* Engaging in 2 or more sessions of strength training exercise per week over a period of at least 3 consecutive months over the past year
* Engaging in aerobic activity at a level that includes competitive events (e.g., marathon, triathlon, running races) over the past year
* Presence of medical conditions or medications that would prohibit participation in an exercise program
* Current use of weight-loss medication
* Documented history of alcohol or substance abuse within the past 12 months
* History of dementia

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Received Dose Intensity (RDI) | Baseline to 26 weeks
  Review of electronic medical records to discern chemotherapy dose received versus prescribed.

SECONDARY OUTCOMES:
Patient-reported chemotoxicities | Baseline to 26 weeks
  Participants will be asked to complete the PRO-CTCAE survey at each chemotherapy cycle. This well-validated survey includes symptoms and adverse events related to chemotherapy. The constructs we will measure include mouth/throat sores, nausea, constipation, diarrhea, neuropathy, concentration, memory, pain, insomnia, and fatigue. A level of 3 or higher will be the threshold for defining a chemotoxicity (yes/no).
Measure of hematologic chemotoxicity - Hematocrit | Baseline to 26 weeks
  Review of medical record to abstract hematocrit values (% of red blood cells in blood).
Measure of hematologic chemotoxicity- White blood cell count | Baseline to 26 weeks
  Review of medical record to abstract white blood cell count.
Measure of hematologic chemotoxicity - Platelet count | Baseline to 26 weeks
  Review of medical record to abstract platelet count.
Measure of hematologic chemotoxicity - Neutrophil count | Baseline to 26 weeks
  Review of medical record to abstract neutrophil count.
Accelerometry | Baseline to 26 weeks
  Physical activity will be measured objectively using Actigraph accelerometry. Accelerometer data will include estimated average metabolic equivalents expended daily and in hours/week as well as time in sedentary, low, moderate and vigorous activity.
Morgenstern Physical Activity Questionnaire (PAQ-M) | Baseline to 26 weeks
  Self-reported physical activity will be measured at baseline and end-of-study using the Morgenstern Physical Activity Questionnaire (PAQ-M), which has been used to reliably capture recreational, occupational and household activity in sedentary adults.
Diet | Baseline to 26 weeks
  Dietary intake will be estimated using repeat administrations of the self-reported, validated Arizona Food Frequency Questionnaire. This questionnaire has been used extensively in large dietary intervention trials among cancer survivors. The instrument will be completed by patients during baseline and end of chemotherapy, reflecting on previous 4 weeks of usual dietary intake.
Strength | Baseline to 26 weeks
  Participants will undergo 10 Repetition Submaximal Strength Testing at baseline and follow-up, collected by the site-based exercise trainer, using a standardized protocol.
MOS SF-36 Questionnaire | Baseline to 26 weeks
  General health-related quality of life (including vitality) will be assessed at baseline and end-of-study using the well-validated MOS SF-36 survey.
Pittsburgh Sleep Quality Index (PSQI) | Baseline to 26 weeks
  Sleep will be assessed at baseline and end-of-study using the PSQI, which is a widely used measure of subjective sleep disturbance; its validity and reliability have been established in various clinical populations, including patients with cancer.
Anthropometric measure - height | Baseline to 26 weeks
  Measure of participant height in centimeters.
Anthropometric measure - weight | Baseline to 26 weeks
  Measure of participant weight in centimeters.
Anthropometric measure - waist circumference | Baseline to 26 weeks
  Measure of participant waist circumference in centimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Schmitz (contact), PhD, MPH, Principal Investigator — University of Pittsburgh; Jennifer Ligibel, MD, Principal Investigator — Dana-Farber Cancer Institute; Nathan Berger, MD, Principal Investigator — Case Western Reserve University/University Hospitals Cleveland
Locations (3):
- United States (3):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Case Western Reserve University/University Hospitals Cleveland, Cleveland, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu